CLINICAL TRIAL: NCT02115490
Title: The Effect of Orally Administered Bisphosphonates in the Treatment of Osteoporosis on the Alveolar Bone Using Panoramic and Cone-Beam CT Imaging: A Case-control Study
Brief Title: Bisphosphonates Effects On Alveolar Bone Among Osteoporotic Women
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-OraMed-01-2014
Record Dates: First submitted 2014-04-11; First posted 2014-04-16 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Osteoporosis
Keywords: Alveolar bone; Bisphosphonates; Cone-beam CT; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Diphosphonates

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Osteoporosis_with_Bisphosphonates: This group of patients are taking Bisphosphonates orally in their treatment
  Interventions: Drug: Bisphosphonates
- Osteoporosis-without-Bisphosphonates: This group of patients has not taken Bisphosphonates in the course of treatment

INTERVENTIONS:
Drug: Bisphosphonates
  Groups: Osteoporosis_with_Bisphosphonates

SUMMARY:
Osteoporosis is a public health problem. It is a skeletal disease being treated by Bisphosphonates as the first choice medication. The effects of these drugs were investigated for periodontal disease treatment both locally and systemically. However, it is very important to know their indirect effects on alveolar bone (i.e. their effects when used for treating osteoporosis). So, in this study, alternations that involve the alveolar bone when osteoporotic women use bisphosphonates will be studied radiologically using cone-beam CT and digital panoramic radiography. The goal is to provide dentists with information about changes in the characterization of the alveolar bone among these women. This is important for both periodontology and implantology. Maxillary and mandibular bone structural characterization among osteoporotic women had not been studied before. Furthermore, in an opposite direction, dental radiographs may aid in detecting osteoporosis.

Osteoporotic women, under bisphosphonates therapy or not, will be invited to participate in this study. In addition, osteopenic and normal women regarding bone fragility will be included too, for comparison purposes. Panoramic radiographs will be taken. In addition, women under bisphosphonates for 6 months or more will be scanned by Cone -beam CT as it can give an idea about bone histomorphometry with a low radiation dose.

DETAILED DESCRIPTION:
Osteoporosis is a skeletal disease characterized by a low bone mass, deterioration of the bone structure and an increased risk of bone fracture. Although jaws are not at risk of fracture, they revealed changes due to the disease. Bisphosphonates are the most common medical therapy for osteoporosis as they improve bone structure and reduce its absorption. From a periodontal point of view, it was suggested as an adjunctive therapy for periodontal bone loss. Controversy exists regarding their effects, however. In addition, their effects on the periodontal status and jaw bones are unknown when these drugs are prescribed for treating osteoporosis, i.e. not for periodontal purposes. It is also unknown whether their effects on alveolar bone, if any, can be detected by simple radiographs (such as panoramic radiographs) or required advanced techniques (e.g. Cone-beam CT).

In this study, their effects on alveolar bone are going to be evaluated using panoramic radiography and Cone-beam CT, as well as the clinical parameters of periodontal diseases. Cone-beam CT will also offer a way to compare bone histomorphometry of the jaws between groups. Bisphosphonates will be prescribed by physicians of osteoporotic women. The investigators will not interfere drug administration at all. Thus, the investigators can test their indirect effect on jaw bones. Osteoporotic women, who used bisphosphonates for 6 months minimum, will be invited to participate in this investigation. In addition, women with osteoporosis who are not under one of the bisphosphonates will be invited too, as a control. Control group will also include a number of osteopenic and normal women for comparison purposes, as these medications are not indicated for them. Women should be free of bone diseases other than osteoporosis or osteopenia.

On panoramic radiographs, radiographic bone density and mandibular cortical index will be assessed. Aluminum step-wedge will be used with panoramic radiography as it offers more accurate density measurements. In Cone-beam CT, radiographic density, apparent bone histomorphometric analysis and radiographic parameters of the periodontal disease will be assessed. Clinical measurements of periodontal disease will be recorded for two purposes. First, to adjust for the confounding factor (periodontal disease) when evaluating the trabecular bone between groups. Second, to test if using these drugs improve the periodontal status as their benefits are still controversial.

ELIGIBILITY:
Inclusion Criteria:

* Women with osteoporosis who already use bisphosphonates.
* Women with osteoporosis who are not under bisphosphonates yet, or are not indicated for such therapy.
* Women with osteopenia either using or not bisphosphonates.

Exclusion Criteria:

* Women with bone diseases other than osteoporosis or osteopenia

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who were referred to perform Dual Energy X-Ray Absorptiometry (DXA) examination will be invited to participate in this study if they were diagnosed with osteoporosis. They may be under bisphosphonates or not. They will be met in Alassd and Almowsat University-Hospitals where DXA is available. If they meet inclusion criteria, mentioned below, they will be invited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
3D-based Alveolar bone radiographic density | One-time assessment; once the woman is scanned by CBCT
  Bone radiographic density will be assessed using special software of cone beam CT

SECONDARY OUTCOMES:
Alveolar bone histomorphometry | One-time assessment; once the patient is scanned by CBCT
  Bone histomorphometry will be assessed using special software used primarily with Micro-CT scans
2D-based Alveolar bone radiographic density | One-time assessment; once the patient is radiographed
  This will be assessed using conventional panoramic radiographs
Periodontal Disease Index (PDI) | One-time assessment in the day of performing the X-ray imaging

CONTACTS AND LOCATIONS:
Overall Officials: Imad Barngkgei, DDS MSc, Principal Investigator — PhD student, Department of Oral Medicine, University of Damascus Dental School, Damascus; Iyad Al-Haffar, DDS MSc PhD, Study Director — Associate Professor of Oral Medicine, Department of Oral Medicine, University of Damascus Dental School, Damascus; Razan Khattab, DDS MSc PhD, Study Director — Professor of Periodontology, Department of Periodontology, University of Damascus Dental School, Damascus, SYRIA
Locations (1):
- University of Damascus Dental School, Damascus, Syrian Arab Republic, Syria

REFERENCES:
- [Background] NIH Consensus Development Panel on Osteoporosis Prevention, Diagnosis, and Therapy, March 7-29, 2000: highlights of the conference. South Med J. 2001 Jun;94(6):569-73. No abstract available. PMID 11440324
- [Background] Darcey J, Devlin H, Lai D, Walsh T, Southern H, Marjanovic E, Horner K. An observational study to assess the association between osteoporosis and periodontal disease. Br Dent J. 2013 Dec;215(12):617-621. doi: 10.1038/sj.bdj.2013.1191. PMID 24357765
- [Background] Devlin H. Identification of the risk for osteoporosis in dental patients. Dent Clin North Am. 2012 Oct;56(4):847-61. doi: 10.1016/j.cden.2012.07.010. Epub 2012 Aug 13. PMID 23017555
- [Background] Doube M, Klosowski MM, Arganda-Carreras I, Cordelieres FP, Dougherty RP, Jackson JS, Schmid B, Hutchinson JR, Shefelbine SJ. BoneJ: Free and extensible bone image analysis in ImageJ. Bone. 2010 Dec;47(6):1076-9. doi: 10.1016/j.bone.2010.08.023. Epub 2010 Sep 15. PMID 20817052
- [Background] Ho JT, Wu J, Huang HL, Chen MY, Fuh LJ, Hsu JT. Trabecular bone structural parameters evaluated using dental cone-beam computed tomography: cellular synthetic bones. Biomed Eng Online. 2013 Nov 9;12:115. doi: 10.1186/1475-925X-12-115. PMID 24207062
- [Background] Jeffcoat MK, Cizza G, Shih WJ, Genco R, Lombardi A. Efficacy of bisphosphonates for the control of alveolar bone loss in periodontitis. J Int Acad Periodontol. 2007 Jul;9(3):70-6. PMID 17715838
- [Background] Kalsi R, Vandana KL, Prakash S. Effect of local drug delivery in chronic periodontitis patients: A meta-analysis. J Indian Soc Periodontol. 2011 Oct;15(4):304-9. doi: 10.4103/0972-124X.92559. PMID 22368351
- [Background] Karaguzel G, Holick MF. Diagnosis and treatment of osteopenia. Rev Endocr Metab Disord. 2010 Dec;11(4):237-51. doi: 10.1007/s11154-010-9154-0. PMID 21234807
- [Background] Koh KJ, Kim KA. Utility of the computed tomography indices on cone beam computed tomography images in the diagnosis of osteoporosis in women. Imaging Sci Dent. 2011 Sep;41(3):101-6. doi: 10.5624/isd.2011.41.3.101. Epub 2011 Sep 15. PMID 22010066